CLINICAL TRIAL: NCT03062826
Title: A Prospective, Multi-center, Optical Coherence Tomography Guided Reperfusion Strategy in Patients With STEMI (EROSION II)
Brief Title: EROSION II: OCT Guided PPCI in STEMI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Harbin Medical University (Other)
Collaborators: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry); Beijing Luhe Hospital (Other); The First Hospital of Jilin University (Other); China-Japan Union Hospital, Jilin University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shanxi Cardiovascular Hospital (Other); Second Hospital of Shanxi Medical University (Other); Hebei General Hospital (Other); General Hospital of Ningxia Medical University (Other); Sichuan Provincial People's Hospital (Other); Affiliated Hospital of Jiangsu University (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); Shenzhen Sun Yat-sen Cardiovascular Hospital (Other); LanZhou University (Other); Sir Run Run Shaw Hospital (Other); Wuhan Asia Heart Hospital (Other)
Responsible Party: Principal Investigator, Yu Bo, Director, The Second Affiliated Hospital of Harbin Medical University
Other Study IDs: HMUOCT-EROSIONII
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: Optical Coherence Tomography; ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Aspirin; Ticagrelor; Clopidogrel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be obtained from artery sheath or coronary artery by aspiration catheter during the PCI procedure in selected sites, and will be stored at -80°C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with STEMI treated medically: Drug: dual antiplatelet therapy (aspirin + ticagrelor or aspirin + clopidogrel) for at least 12 months.
  Interventions: Drug: dual antiplatelet therapy (aspirin + ticagrelor or aspirin + clopidogrel)

INTERVENTIONS:
Drug: dual antiplatelet therapy (aspirin + ticagrelor or aspirin + clopidogrel) — Patients who met the inclusion criteria will be treated with dual antiplatelet therapy (aspirin + ticagrelor or aspirin + clopidogrel).

SUMMARY:
This protocol describes a prospective, multi-center study intended to test the hypothesis that patients with STEMI caused by plaque rupture or plaque erosion without obstructive stenosis (diameter stenosis <70%) can be stabilized by effective antithrombotic treatment without stent implantation, thereby avoiding both early and late complications related to percutaneous coronary intervention (PCI) with stent implantation. All the patients will be followed by intracoronary OCT and physiological assessment at 1-month and 12-month follow-up.

DETAILED DESCRIPTION:
EROSION (Effective anti-thrombotic therapy without stenting: intravascular optical coherence tomography-based management in plaque erosion) study, a single-center, uncontrolled, prospective, proof-of concept study, showed that for patients with ACS caused by non-obstructive plaque erosion, conservative treatment with anti-thrombotic therapy without stenting may be an option. However, it is unknown whether plaque rupture with large lumen area and non-obstructive stenosis can be treated medically without stenting. EROSION II study is a prospective, multi-center, observational study to test the hypothesis that patients with STEMI caused by plaque rupture or plaque erosion without obstructive stenosis (diameter stenosis <70% by visual assessment) can be stabilized and healed by effective antithrombotic treatment without stent implantation. Patients presenting with STEMI within 24 hours from the onset of ischemic symptoms will be included for screening. Thrombus aspiration will be performed in patients with large thrombus burden and TIMI flow grade less than 2 to restore blood flow. OCT will be performed after antegrade blood flow restored to assess the underlying mechanism of culprit lesion including plaque rupture, plaque erosion, calcified nodule, spontaneous coronary artery dissection, and other uncommon reasons. OCT imaging of non-culprit vessels will be performed if feasible. Patients caused by plaque erosion or plaque rupture with minimal lumen area > 1.6mm2 or non-obstructive stenosis (diameter stenosis <70% by visual assessment) will be treated medically only with dual anti-platelet therapy for 12 months after discharge.

Serial OCT examination will be performed at 1-month and 12-month follow-up to assess the healing of original culprit lesion. Physiological assessment (either wire-based FFR or angio-based FFR) will also be performed to assess the hemodynamic function of culprit lesion. The primary endpoint is the reduction of thrombus burden assessed by OCT at 1-month follow-up. Presence of recurrent ischemia symptoms or positive FFR value are the indications for target lesion revascularization. Patients will be followed by phone calls by study coordinators or clinical visit at 1 month, 3 months, 6 months, 9 months and 12 months. Major cardiovascular adverse events (MACE) will be collected in all patients throughout the whole follow-up period. MACE is a composite of cardiac death, recurrent myocardial infarction, stroke, target lesion revascularization, major bleeding and unstable angina-induced rehospitalization.

Patients who do not meet the criteria after OCT imaging will be enrolled in registry cohort.

Blood sample will be obtained from artery sheath or coronary artery by aspiration catheter during the PCI procedure in selected sites. Blood samples will be stored at -80°C for potential biomarker test and multi-omics analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women >18 years of age and < 75 years of age.
* Patients undergo cardiac catheterization for STEMI. STEMI will be defined as continuous chest pain for >30 minutes, arrival at the hospital within 24 hours from chest pain onset, ST-segment elevation >0.1 mV in at least two contiguous leads, or new left bundle-branch block on the 12-lead electrocardiogram (ECG), and elevated cardiac markers (troponin T/I or creatine kinase-MB).
* Culprit lesion located in a native coronary artery.
* TIMI flow grade 3 and diameter stenosis < 70% by visual assessment on angiogram or MLA > 1.6mm2.
* Plaque erosion and rupture defined by OCT.
* Patients able to provide written informed consent.

Exclusion Criteria:

* Left ventricular ejection fraction < 30%.
* Lesions in LM, ostial LAD or RCA (defined as within 3 mm of the aorto-ostium).
* Long lesions, tortuous lesions and angulated lesions.
* More than 2 vessels with severe lesions.
* Massive residual thrombus after the thrombus aspiration.
* With the history of cardiopulmonary resuscitation (CPR), acute pulmonary edema and cardiac shock on the attacks.
* Life expectancy < 1 year.
* Contraindication to the contrast media.
* Creatinine level > 2.0 mg/dL or end-stage kidney disease.
* Serious liver dysfunction.
* Patients with hemodynamic or electrical instability (including shock).
* Any contraindication against the use of ticagrelor.
* Investigator considers the patient is not suitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is STEMI patients who undergo primary cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of thrombus burden assessed by OCT | 30 days
  The efficacy will be assessed by 50% reduction in thrombus burden by OCT at 1 month.

SECONDARY OUTCOMES:
Major cardiovascular adverse events | 1, 3, 6, 9, 12 months after PCI
  In patients treated conservatively, the safety objectives are to evaluate the occurrence of any adverse events during 1, 3, 6, 9, 12 months follow up (re-infarction, re-hospitalization due to unstable angina, revascularization by PCI or CABG, cardiac death, stroke, and major bleeding).
Major cardiovascular adverse events | 1 and 12 months after PCI
  compare the difference of clinical outcome in patients with plaque rupture and erosion.
Effective flow area increase | 1 and 12 months after PCI
  Effective flow area increase
Fractional flow reserve | 1 and 12 months after PCI
  either wire-based FFR or angio-based FFR

CONTACTS AND LOCATIONS:
Overall Officials: Bo YU, MD, PhD, Study Chair — The Second Affiliated Hospital of Harbin Medical University
Locations (16):
- China (16):
  - Beijing Luhe Hospital, Beijing, Beijing Municipality
  - Xiamen Cardiovascular Hospital, Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Shenzhen Sun Yat-sen Cardiovascular Hospital, Shenzhen, Guangzhou
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Shenyang
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2020